CLINICAL TRIAL: NCT05058287
Title: Topical Epidural Steroid Usage in Patients Undergoing Posterior Lumbar Decompression: A Randomized Control Trial
Brief Title: Lumbar Steroid Use in Patients Undergoing Posterior Lumbar Decompression
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-0041
Record Dates: First submitted 2021-08-09; First posted 2021-09-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-01

CONDITIONS: Opioid Use; Lumbar Spinal Stenosis; Pain, Postoperative; Pain, Back
MeSH Terms: conditions — Spinal Stenosis; Pain, Postoperative; Back Pain | interventions — Methylprednisolone Acetate; Suspensions; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Topical Steroid (Experimental)
  Interventions: Drug: Depo-Medrol 40Mg/Ml Suspension for Injection
- Group 2: Topical Normal Saline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Depo-Medrol 40Mg/Ml Suspension for Injection — 40mg Depo-Medrol mixed with hemostatic matrix
  Arms: Group 1: Topical Steroid
Drug: Placebo — 1 mL of sterile normal saline mixed with hemostatic matrix
  Arms: Group 2: Topical Normal Saline

SUMMARY:
This study seeks to evaluate the impact of intra-operative topical epidural steroid usage in patients undergoing 1-2 level lumbar laminectomy. The study will examine post-operative opioid usage, length of stay, return to work, and patient reported outcomes following these procedures.

DETAILED DESCRIPTION:
This is a randomized controlled trial seeking to evaluate the impact of intra-operative topical epidural steroid usage in patients undergoing 1- to 2- level lumbar laminectomies. Subjects enrolled in this study will be randomized to one of two treatments: either 40 mg Depo-Medrol or 1 mL of sterile normal saline will be applied to the surgical wound prior to closure. The study will examine post-operative opioid usage, length of stay, return to work, and patient reported outcomes following these procedures. Subjects will be assessed pre-operatively, while admitted for surgery, and postoperatively daily for two weeks, then again at 1- and 3- months.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo 1 to 2 level laminectomy
* Between the ages of 18-85

Exclusion Criteria:

* Minimally invasive surgery
* Prior daily opioid usage within 6 months.
* Use of concomitant procedures such as spinal fusion, revision procedure at the same level.
* History of a chronic pain syndrome, uncontrolled diabetes defined as A1C > 6.5, immunocompromised condition such as active cancer treatment, history of transplant, benign prostatic hyperplasia or history of urinary retention, and other conditions which require chronic steroid therapy or immunosuppressants.
* Non-English speakers
* Patients allergic to Depo-Medrol and/or glucocorticoids, or other steroids

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid use total [Both Groups] | In hospital, pre-discharge
  Number & dose of opioid taken converted to oral morphine equivalents post-operatively in hospital
Opioid use total [Both Groups] | Every day for 14 days post- discharge
  Number & dose of opioid taken converted to oral morphine equivalents post-operatively post-discharge
Opioid consumption [Both Groups] | 6-Week Post-Op
  Is participant still taking post-op opioids
Opioid consumption [Both Groups] | 3-Months Post-Op
  Is participant still taking post-op opioids

SECONDARY OUTCOMES:
Numeric Rating Pain Scale [Both Groups] | pre-operative
  Baseline pain as measured through the NRS 0: None; 1,2,3: Mild; 4,5,6: Moderate; 7,8,9,10: Severe
Numeric Rating Pain Scale [Both Groups] | every day for 14 days post-op
  Change in baseline pain as measured through the NRS Scale: 0-10 0: None; 1,2,3: Mild; 4,5,6: Moderate; 7,8,9,10: Severe;
Numeric Rating Pain Scale [Both Groups] | 6-week
  Change in baseline pain as measured through the NRS Scale: 0-10 0: None; 1,2,3: Mild; 4,5,6: Moderate; 7,8,9,10: Severe
Numeric Rating Pain Scale [Both Groups] | 3-month follow up
  Change in baseline pain as measured through the NRS Scale: 0-10 0: None; 1,2,3: Mild; 4,5,6: Moderate; 7,8,9,10: Severe
Veterans Rand 12-Item Health Survey [Both Groups] | pre-operative
  Baseline pain as measured through VR-12
Veterans Rand 12-Item Health Survey [Both Groups] | 2 week post-op
  Change in baseline pain as measured through VR-12
Veterans Rand 12-Item Health Survey [Both Groups] | 6 week post-op
  Change in baseline pain as measured through VR-12
Veterans Rand 12-Item Health Survey [Both Groups] | 3 month post-op
  Change in baseline pain as measured through VR-12
Oswestry Low Back Pain Disability Questionnaire [Both Groups] | pre-operative
  Baseline pain as measured through ODI
Oswestry Low Back Pain Disability Questionnaire [Both Groups] | 2 week
  Change in baseline pain as measured through ODI
Oswestry Low Back Pain Disability Questionnaire [Both Groups] | 6 week
  Change in baseline pain as measured through ODI
Oswestry Low Back Pain Disability Questionnaire [Both Groups] | 3 month follow up
  Change in baseline pain as measured through ODI
Return to Work [Both Groups] | 2 week
  Date participant returned to work
Return to Work [Both Groups] | 6 week
  Date participant returned to work
Return to Work [Both Groups] | 3 month follow up
  Date participant returned to work
Medical Complications [Both Groups] | 2 week
  Any medical complications
Medical Complications [Both Groups] | 6 week
  Any medical complications
Medical Complications [Both Groups] | 3 month follow up
  Any medical complications
Re-admissions [Both Groups] | 2 Week
  Any re-admissions
Re-admissions [Both Groups] | 6 Week
  Any re-admissions
Re-admissions [Both Groups] | 3 Month
  Any re-admissions

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified data after all study related activities are completed.
Supporting Information: CSR
Time Frame: We plan to share de-identified data after all study related activities are completed for a minimum of 1 year.
Access Criteria: The data will be posted through PRS